CLINICAL TRIAL: NCT06960876
Title: Comparative Effects of Therapeutic Ultrasound and Sinus Massage in Chronic Rhinosinusitis: a Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/68
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Chronic Rhinosinusitis (CRS)
Keywords: CHRONIC RHINOSINUSITIS; Therapeutic ultrasound; sinus massage
MeSH Terms: interventions — Ultrasonic Therapy; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): All three groups will continue their prescribed steam protocol and medications by the ENT specialist Group A will additionally receive a therapeutic Ultrasound over the maxillary sinus
  Interventions: Procedure: Therapeutic Ultrasound
- Group B (Experimental): All three groups will continue their prescribed steam protocol and medications by the ENT specialist Group B will additionally receive, sinus massage (pressure & milking)
  Interventions: Procedure: Sinus Massage
- Group C (Active Comparator): All three groups will continue their prescribed steam protocol and medications by the ENT specialist Group C will not receive any other adjunct physical therapy treatment (control group)
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Therapeutic Ultrasound — All three groups will continue their prescribed steam protocol and medications by the ENT specialist. This Group will additionally receive a therapeutic Ultrasound over the maxillary sinus.
  Arms: Group A
Procedure: Sinus Massage — All three groups will continue their prescribed steam protocol and medications by the ENT specialist. This group will additionally receive, sinus massage (pressure & milking)
  Arms: Group B
Procedure: Control group — All three groups will continue their prescribed steam protocol and medications by the ENT specialist. This group will not receive any other adjunct physical therapy treatment (control group)
  Arms: Group C

SUMMARY:
This is a randomized controlled trial. Previous studies show that both therapeutic ultrasound and sinus massage techniques have significant results in Chronic Rhinosinustis (CRS).

However, there is no comparative study carried out between these two to show which technique has more effects in CRS.

This study will determine their comparative effects on:

1. Pain measured on Numerical pain rating scale
2. Sinonasal symptoms measured on sino-nasal outcome test questionaire
3. Quality of life measured on rhinosinusitis disability index (RSDI)
4. Nasal inspiratory airflow measured on peak nasal inspiratory flow meter. Participants of chronic rhinosinusitis will be selected according to the diagnostic criteria of American Academy of Otolaryngology-Head and Neck Surgery Foundation (AAO-HNSF) and will be randomly allocated into three groups. All three group will continue to receive medical intervention. Additionally one group will receive therapeutic ultrasound while other group will receive sinus massage. Whereas third group will be control group and won't receive any additional treatment.

Data will be collected at Foundation University College of Physical Therapy and Fauji Foundation Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years
* Both gender
* Diagnosed patients of chronic rhinosinusitis referred by an ENT specialist
* According to the AAO-HNS, patients are diagnosed with CRS if they had:
* Two or more major symptoms for ≥12 weeks. Or
* one major symptom with two minor symptoms for ≥12 weeks (19) Major clinical symptoms
* Pain or pressure on the face
* Nasal congestion
* Mucopurulent rhinorrhea either anteriorly, posteriorly, or both
* Hyposmia/anosmia Minor clinical symptoms
* Headache
* Fever
* Pain in the dental area
* Halitosis
* Pain or pressure on the ear
* Cough

Exclusion Criteria:

* Nasal polyps
* Current Medical conditions in which ultrasound is contraindicated (20)
* Facial metal implants
* Face or head tumor/cyst/malignancy
* Deteriorated cognitive level
* Previous surgery on the nose
* Facial bone fracture
* Reduced heat perception
* Ischemic tissues
* Skin allergies/lesions to the face

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Pain level | 4 weeks
  The numeric pain rating scale will be used. The participants rate their pain from 0-10.
  Scoring: 0 shows no pain, whereas 10 represents the worst pain.
sino-nasal symptoms | 6 weeks
  Sino-nasal outcome test questionnaire for assessing sino-nasal symptoms The SNOT-22 is a 22-item treatment outcome measure designed for people with chronic sinonasal conditions. The SNOT-22 has been evaluated and is based on a Likert scale. Scoring: 0="No problem", 1="Very mild problem", 2="Mild or slight problem", 3="Moderate problem", 4="Severe problem", and 5="Problem as bad as it can be." Higher scores on SNOT-22 survey items indicate worse patient function or more severe symptoms (total score range: 0-110)
health-related quality of life (HRQL) in rhinosinusitis | 6 weeks
  Rhino Sinusitis Disability Index (RSDI) for measuring health-related quality of life (HRQL) in rhinosinusitis The purpose of this scale is to identify difficulties experienced due to nose or sinus problems. The Rhinosinusitis Disability Index (RSDI) has a total score range of 0-120 and consists of 30 items.
nasal inspiratory flow rate | 6 weeks
  Peak nasal inspiratory flow meter to evaluate nasal inspiratory flow rate during maximal inspiration It works when a patient inhales through the nose causing air to be drawn through the meter, a cursor moves along the scale to indicate the speed of inhalation. The flow rate achieved can be noted by checking the position of the cursor against the calibrated scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan